CLINICAL TRIAL: NCT04952766
Title: Study Evaluating SARS-CoV-2 (COVID-19) Humoral Response After BNT162b2 Vaccine in Immunocompromised Adults Compared to Healthy Adults
Acronym: EREVA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre Hospitalier Régional d'Orléans (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHRO-2021-04
Record Dates: First submitted 2021-06-16; First posted 2021-07-07 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Kidney Transplant; Myeloma; Cancer; Hematologic Malignancy; Multiple Sclerosis; Hypergammaglobulinemia; Malignant Tumor; Hiv; Diabetes Type 2
Keywords: SARS-CoV-2; BNT162b2 vaccine; antibody; neutralization; mucosa; immunocompromised; healthy subject
MeSH Terms: conditions — Neoplasms, Plasma Cell; Neoplasms; Hematologic Neoplasms; Multiple Sclerosis; Hypergammaglobulinemia; Acquired Immunodeficiency Syndrome; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: All participants wil have at each of the 4 visits (for patients starting at month 1) or 5 visits (for patients starting at month 0):
  1. a venipuncture sample of 2 dry tubes of 7 mL (less than 30 mL in total) to make up 3 aliquots and
  2. a nasopharyngeal swab (optional). The aliquots of serum / plasma and the nasopharyngeal swab will be stored at -80°C until sent to the Pasteur Institute.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- immunocompromised and healthy subjects (Other): Immunocompromised subjects and healthy subjects groups will have collection of biological samples (blood with/without nasopharyngeal swabs) at Month-0, -1, -2, -3, -6, with associated data for the study of the kinetics of antibodies anti COVID-19.
  Biological samples :
  * Serum and plasma from each participant for the purpose of performing the SARS-CoV-2 serologic tests
  * Nasopharyngeal samples (not mandatory)
  Associated data :
  * Demographic data
  * Description of clinical manifestations related to vaccination
  * Description of clinical manifestations related to SARS-CoV-2 infection, if any Blood Fractioning
  * Serum and plasma aliquoted and stored under 250, 500 and 1000 µL (at -80°C)
  Interventions: Biological: Biological samples

INTERVENTIONS:
Biological: Biological samples — Immunocompromised subjects and healthy subjects groups will have collection of biological samples (blood with/without nasopharyngeal swabs) at Month-0, -1, -2, -3, -6, with associated data for the study of the kinetics of antibodies anti COVID-19.
  Biological samples :
  * Serum and plasma from each participant for the purpose of performing the SARS-CoV-2 serologic tests
  * Nasopharyngeal samples (not mandatory)
  Associated data :
  * Demographic data
  * Description of clinical manifestations related to vaccination
  * Description of clinical manifestations related to SARS-CoV-2 infection, if any Blood Fractioning
  * Serum and plasma aliquoted and stored under 250, 500 and 1000 µL (at -80°C)

SUMMARY:
The primary endpoint of this study is to compare the humoral response (titre and neutralizing capacity of induced antibodies) against SARS-CoV-2 following vaccination with BNT162b2 (Pfizer BioNTech) in immunocompromised persons, in comparison to healthy subject. Secondary objectives are to evaluate the humoral response in the nasal mucosa, and the capacity of antibodies to neutralize emerging variants of concerns and to prevent COVID-19.

DETAILED DESCRIPTION:
The serious, even fatal, forms of COVID-19 preferentially affect elderly and fragile subjects. Among these populations at risk, people who are immunocompromised (either by a disease and / or its treatment) have a theoretical risk of responding less well to a preventive vaccination.

The main objective of this study aims to compare the vaccine response of immunocompromised people with healthy subjects (non-immunocompromised), i.e. to assess the serum humoral response (titre and neutralizing capacity of the antibodies induced) following vaccination with ComirnatyTM (i.e. BNT162b2, an anti-SARS-CoV-2 vaccine from Pfizer BioNTech) in immunocompromised persons in comparison to healthy subjects (non-immunocompromised).

Secondary objectives are as follows:

* To evaluate the antibody response in the nasal mucosa (titre and neutralizing capacity of the antibodies induced, collected by means of a nasopharyngeal swab) following vaccination with ComirnatyTM in immunocompromised people as compared to healthy subjects (vaccinated either with two doses of ComirnatyTM or, in a subgroup, with one dose of Astra Zeneca's VaxzeriaTM followed by one dose of ComirnatyTM).
* Evaluate the serum and mucosal antibody response (titre and neutralizing capacity of the antibodies induced) against emerging strains of SARS-CoV-2 (so-called Alpha, Beta, Gamma, Delta strains).
* Evaluate the post-vaccination clinical protection against the risk of COVID-19 infection (incident cases after vaccination).

ELIGIBILITY:
Inclusion Criteria:

* Adult volunteers to be vaccinated with the ComirnatyTM vaccine and to participate in the study, belonging to one of the following groups:

  * Group of immunocompromised (15 participants per immunosuppression subgroup):

    * Kidney transplant
    * Extracorporeal dialysis
    * Solid cancer under chemotherapy and / or radiotherapy
    * Myeloma under chemotherapy
    * Hematologic malignancies under chemotherapy
    * Diseases treated with anti CD20 (or patients not treated at the time of the vaccine but who will be immediately after)
    * Multiple sclerosis under anti CD20 (or patients not treated at the time of the vaccine but who will be immediately after)
    * Common variable immune deficiency or other causes of severe hypogammaglobulinemia requiring chronic treatment with polyvalent immunoglobulin
    * Malignant tumor under anti-PD1 or anti-PDL1
    * People living with HIV
    * Complicated type 2 diabetes (with micro and / or macroangiopathy)
  * Group of non-immunocompromised subjects (controls, n = 75)

    * 60 people vaccinated with the ComirnatyTM
    * 15 people vaccinated with Astra Zeneca's VaxzevriaTM for the first dose

Exclusion Criteria:

* Minors
* Pregnant or breastfeeding women
* Persons under tutorship or curatorship
* Protected adults
* Person under legal protection
* Person not affiliated to a social security scheme
* People with a contraindication to receiving the ComirnatyTM vaccine
* People who have already been vaccinated against SARS-CoV-2

Note: a history of COVID-19 (> at 3 months) is not a contraindication to vaccination and is therefore not a criterion for non-inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2021-03-26 (Actual); Primary Completion 2022-02-06 (Actual); Study Completion 2022-02-06 (Actual)

PRIMARY OUTCOMES:
Protective humoral response after vaccination | Month 2
  Proportion of immunocompromised persons with neutralizing activity against the classic "Wuhan" strain of SARS-CoV-2 compared to the proportion obtained in healthy subjects.

SECONDARY OUTCOMES:
Mucosal neutralization capacity against wild-type and emerging variants of concern (VOC) | Month 0
  Proportion of immunocompromised people with neutralizing activity in the nasal mucosa against the classic "Wuhan" strain of SARS-CoV-2 compared to the proportion obtained in healthy subjects.
Mucosal neutralization capacity against wild-type and emerging variants of concern (VOC) | Month 1
  Proportion of immunocompromised people with neutralizing activity in the nasal mucosa against the classic "Wuhan" strain of SARS-CoV-2 one month after the second dose of the vaccine, compared to the proportion obtained in healthy subjects.
Mucosal neutralization capacity against wild-type and emerging variants of concern (VOC) | Month 2
  Proportion of immunocompromised people with neutralizing activity in the nasal mucosa against the classic "Wuhan" strain of SARS-CoV-2 compared to the proportion obtained in healthy subjects.
Mucosal neutralization capacity against wild-type and emerging variants of concern (VOC) | Month 3
  Proportion of immunocompromised people with neutralizing activity in the nasal mucosa against the classic "Wuhan" strain of SARS-CoV-2 compared to the proportion obtained in healthy subjects.
Mucosal neutralization capacity against wild-type and emerging variants of concern (VOC) | Month 6
  Proportion of immunocompromised people with neutralizing activity in the nasal mucosa against the classic "Wuhan" strain of SARS-CoV-2 compared to the proportion obtained in healthy subjects.
Serum and nasal neutralization capacity against wild-type and emerging variants of concern (VOC) | Month 0
  Proportion of immunocompromised people with neutralizing activity in the serum and nasal mucosa against emerging strains of SARS-CoV-2 (so-called Alpha, Beta, Gamma, Delta strains)
Serum and nasal neutralization capacity against wild-type and emerging variants of concern (VOC) | Month 1
  Proportion of immunocompromised people with neutralizing activity in the serum and nasal mucosa against emerging strains of SARS-CoV-2 (so-called Alpha, Beta, Gamma, Delta strains)
Serum and nasal neutralization capacity against wild-type and emerging variants of concern (VOC) | Month 2
  Proportion of immunocompromised people with neutralizing activity in the serum and nasal mucosa against emerging strains of SARS-CoV-2 (so-called Alpha, Beta, Gamma, Delta strains)
Serum and nasal neutralization capacity against wild-type and emerging variants of concern (VOC) | Month 3
  Proportion of immunocompromised people with neutralizing activity in the serum and nasal mucosa against emerging strains of SARS-CoV-2 (so-called Alpha, Beta, Gamma, Delta strains)
Serum and nasal neutralization capacity against wild-type and emerging variants of concern (VOC) | Month 6
  Proportion of immunocompromised people with neutralizing activity in the serum and nasal mucosa against emerging strains of SARS-CoV-2 (so-called Alpha, Beta, Gamma, Delta strains)
Clinical protection after vaccination | Month 0
  Proportion of participants developing COVID-19 infection after vaccination
Clinical protection after vaccination | Month 1
  Proportion of participants developing COVID-19 infection after vaccination
Clinical protection after vaccination | Month 2
  Proportion of participants developing COVID-19 infection after vaccination
Clinical protection after vaccination | Month 3
  Proportion of participants developing COVID-19 infection after vaccination
Clinical protection after vaccination | Month 6
  Proportion of participants developing COVID-19 infection after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Aymeric SEVE, Dr, Principal Investigator — CHU Orléans
Locations (1):
- CHU Orléans, Orléans, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grzelak L, Temmam S, Planchais C, Demeret C, Tondeur L, Huon C, Guivel-Benhassine F, Staropoli I, Chazal M, Dufloo J, Planas D, Buchrieser J, Rajah MM, Robinot R, Porrot F, Albert M, Chen KY, Crescenzo-Chaigne B, Donati F, Anna F, Souque P, Gransagne M, Bellalou J, Nowakowski M, Backovic M, Bouadma L, Le Fevre L, Le Hingrat Q, Descamps D, Pourbaix A, Laouenan C, Ghosn J, Yazdanpanah Y, Besombes C, Jolly N, Pellerin-Fernandes S, Cheny O, Ungeheuer MN, Mellon G, Morel P, Rolland S, Rey FA, Behillil S, Enouf V, Lemaitre A, Creach MA, Petres S, Escriou N, Charneau P, Fontanet A, Hoen B, Bruel T, Eloit M, Mouquet H, Schwartz O, van der Werf S. A comparison of four serological assays for detecting anti-SARS-CoV-2 antibodies in human serum samples from different populations. Sci Transl Med. 2020 Sep 2;12(559):eabc3103. doi: 10.1126/scitranslmed.abc3103. Epub 2020 Aug 17. PMID 32817357
- [Background] Planas D, Bruel T, Grzelak L, Guivel-Benhassine F, Staropoli I, Porrot F, Planchais C, Buchrieser J, Rajah MM, Bishop E, Albert M, Donati F, Prot M, Behillil S, Enouf V, Maquart M, Smati-Lafarge M, Varon E, Schortgen F, Yahyaoui L, Gonzalez M, De Seze J, Pere H, Veyer D, Seve A, Simon-Loriere E, Fafi-Kremer S, Stefic K, Mouquet H, Hocqueloux L, van der Werf S, Prazuck T, Schwartz O. Sensitivity of infectious SARS-CoV-2 B.1.1.7 and B.1.351 variants to neutralizing antibodies. Nat Med. 2021 May;27(5):917-924. doi: 10.1038/s41591-021-01318-5. Epub 2021 Mar 26. PMID 33772244